CLINICAL TRIAL: NCT04843865
Title: A Systemic Approach to Study the Traditional Chinese Medicine as an Adjuvant Treatment in Breast Cancer Patients
Brief Title: TCM as an Adjuvant Treatment in Breast Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Yang Mooi Lim, Professor, Universiti Tunku Abdul Rahman
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTAR- 8068/000
Record Dates: First submitted 2021-03-19; First posted 2021-04-14 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Musculoskeletal Pain
Keywords: Chinese herbs; Breast cancer; Aromatase inhibitor-associated musculoskeletal symptoms; Protein profiling; System biology; Syndrome element differentiation
MeSH Terms: conditions — Breast Neoplasms; Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: A quasi-experimental design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chinese Herbs (Experimental): Participants received standardized Chinese Herbs treatment orally twice daily for 1 week.
  Interventions: Dietary Supplement: Chinese Herbs

INTERVENTIONS:
Dietary Supplement: Chinese Herbs — Chinese Herbs

SUMMARY:
Chinese herbs can alleviates the side effects caused by conventional treatment in breast cancer patients and affects the syndrome element differentiation by altering the specific set of proteomes at specific time point of treatment.

DETAILED DESCRIPTION:
The previous studies have reported that adjuvant Chinese herbs therapy can improve the survival of breast cancer patients by alleviating the side effects of conventional treatments. Protein expression determines the phenotype of a patient that contributes to the onset of side effects in breast cancer patients caused by conventional treatment. Chinese herbs treatment will alleviate the treatment-related side effects by altering the protein expression in the patients. Associating changes in protein levels with the onset of side effects caused by conventional treatments could be used to identify clinically relevant diagnostic biomarkers. In addition, a set of proteome that is being expressed at diseased state will exhibit the phenotype that is also correlated to the TCM syndrome differentiation. Hence, this study aims to determine the proteome profile for the syndrome differentiation of breast cancer patients treated with adjuvant Chinese herbs for musculoskeletal pain. A quasi-experimental study with purposive sampling will be conducted on 30 breast cancer patients recruited from Tung Shin hospital. All participants will be invited to complete a structured questionnaire to collect their demographic information, pain score, syndrome element differentiation, quality of life, stress, body constitution and other relevant information, including cancer type, cancer stage, and cancer treatment. The questionnaires will be self-administered either at the outpatient waiting room or in the ward of the study hospital. Blood of the patients will be collected for determination of protein expression, biochemical markers and cytokines. The study is an in-point analysis where 2 time-points of data collection and analysis will be carried out at baseline, and immediate post Chinese herbs treatment. Informed consent will be obtained before participant enrolment according to a clinical trial protocol. Statistical differences for protein expression, biochemical markers, cytokines and mean pain score before and after Chinese herbs treatment will be compared using the paired-sample t test.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women as determined by cessation of menses for at least 1 year or FSH>20 mIU/mL
* Histology confirmed stage 2 to 3 hormone-receptor positive breast cancer patient
* Currently taking letrozole for at least 1 month
* Reported ongoing musculoskeletal pain or stiffness, which started or worsened after initiation of letrozole
* Had a baseline average pain score over the past week on the Brief Pain Inventory Short Form (BPI-SF) of ≥4 points on a scale of 0 to 10.
* Completed all indicated surgery, chemotherapy and radiation therapy
* Agreed to take prescribed Chinese herbs
* No evidence of distant metastasis
* Follow-up for the duration of the study
* No acute disease in the past month
* Able to communicate to practitioner and interviewer
* Willing to give informed consent

Exclusion Criteria:

* Pregnant or nursing woman or woman of childbearing potential without effective method of birth control.
* Patients who default subsequent follow-up/ has irregular follow-up.
* Patients who directly involved in other study at the same time.
* History of non-compliance to medical regime and patients who are unwilling or unable to comply with the protocol.
* Bedridden and/ or cancer metastasis to bone/ lung.
* Concurrent infection requiring intravenous antibiotics
* History of allergy to Chinese herbs
* Had previously received Chinese herbs for their AI-induced musculoskeletal symptoms
* Had received Chinese herbs within one month prior to study entry
* Current use of steroids or narcotics for pain relief within the past 2 weeks
* Subjects with acute onset of a chronic illness or with acute disease in the past month or had pre-existing chronic diseases
* Patients with concomitant severe illness or metastatic disease (poorly controlled hypertension, hypothyroidism, diabetes mellitus, liver diseases, osteoarthritis, rheumatoid arthritis, gout or neuropathic arthropathy, autoimmune or inflammatory joint disease, bone fracture, stroke)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the study (Adherence) | Immediate post 1 week of Chinese Herbs intervention
  The feasibility of the adherence will be determined by the number of sachets of Chinese herbs taken.

SECONDARY OUTCOMES:
Feasibility of the study (Dropout rate) | Immediate post 1 week of Chinese Herbs intervention
  The feasibility will be assessed by dropout rate of the patients.
Change in the pain score | Baseline and immediate post 1 week of Chinese Herbs intervention
  The pain score of breast cancer patients will be assessed by Brief Pain Inventory-Short Form (BPI-SF). BPI-SF is a validated and reliable tool used to assess the severity or intensity of pain on scale ranging from 0 (no pain) to 10 (worst pain imaginable). Higher scores mean a worse outcome.
Change in Syndrome element differentiation | Baseline and immediate post 1 week of Chinese Herbs intervention
  Syndrome Element Differentiation rating scale will be used to determine the syndrome element differentiation of the patients. Syndrome Element Differentiation rating scale can quantify the syndrome elements of this patient based on the clinical manifestations. The quantitative output weight values of syndrome elements are acquired from clinical input data based on the severity and frequency of each sign and symptom. Based on the quantitative output value, the syndrome elements can then be categorized into four levels of health state or severity: normal (<70), mild (≥ 70 to <100), moderate (≥100 to <150), and severe (≥ 150).
Change in quality of life as assessed by WHO-BREF (World Health Organization Quality of Life) | Baseline and immediate post 1 week of Chinese Herbs intervention
  The quality of life will be assessed by the WHO-BREF questionnaire in this study. The WHOQOL-BREF instrument comprises 26 items, measuring the following broad domains: physical health, psychological health, social relationships, and environment, with scores ranging from 0 to 100. The four domain scores denote an individual's perception of the quality of life in each domain. Domain scores are scaled in a positive direction in which higher scores denote a higher quality of life.
  * the minimum and maximum values: 0, 100
  * higher scores mean a better outcome.
Change in stress | Baseline and immediate post 1 week of Chinese Herbs intervention
  The Depression Anxiety Stress Scales (DASS) is a self-report instrument designed to measure the negative emotional states of depression, anxiety and stress. A short version, the DASS 21 scale consists of a list of 21 symptoms with 7 item per scale, each of which is to be rated on a four-point scale of how much you had that symptom in the last week from 'never' to 'most of the time'. In this study, stress will be determined by stress domain of DASS-21 which consists of 7 items.
Change in body constitution assessed by Constitution in Chinese Medicine Questionnaire (CCMQ) | Baseline and immediate post 1 week of Chinese Herbs intervention
  The body constitution will be determined by Constitution in Chinese Medicine Questionnaire (CCMQ). It has 60 items measuring the 9 body constitution types: gentleness, Qi-deficiency, Yang-deficiency, Yin-deficiency, phlegm-wetness, wetness-heat, blood-stasis, Qi-depression, and special diathesis.
  * the minimum and maximum values: 0, 100
  * higher scores mean a worse outcome.
Change in protein expression | Baseline and immediate post 1 week of Chinese Herbs intervention
  The serum proteome will be analyzed by liquid chromatography coupled with tandem mass spectrometry (LC-MS/MS).
Change in Liver Function Test | Baseline and immediate post 1 week of Chinese Herbs intervention
  The liver function of the patients will be determined by measuring the alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase.
Change in CEA (Carcino-Embryonic Antigen) | Baseline and immediate post 1 week of Chinese Herbs intervention
  Change in CEA (Carcino-Embryonic Antigen) will be determined by laboratory examination.
Change in CRP (C-Reactive Protein) | Baseline and immediate post 1 week of Chinese Herbs intervention
  Change in CRP (C-Reactive Protein) will be determined by laboratory examination.
Change in Progesterone | Baseline and immediate post 1 week of Chinese Herbs intervention
  Change in Progesterone will be determined by laboratory examination.
Change in Estradiol | Baseline and immediate post 1 week of Chinese Herbs intervention
  Change in Estradiol will be determined by laboratory examination.
Change in Cytokine levels of serum | Baseline and immediate post 1 week of Chinese Herbs intervention
  The cytokines in serum samples of breast cancer patients will be detected by the Quantibody array, multiplexed sandwich enzyme-linked immunosorbent assay (ELISA) based quantitative array platform (Genomax technology) for quantitative measurement of cytokines in human serum. The unit of measurement for the cytokines is the same.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Mooi Lim, Principal Investigator — Universiti Tunku Abdul Rahman (UTAR)
Locations (1):
- Tung Shin Hospital, Bukit Bintang, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nie J, Zhao C, Deng LI, Chen J, Yu B, Wu X, Pang P, Chen X. Efficacy of traditional Chinese medicine in treating cancer. Biomed Rep. 2016 Jan;4(1):3-14. doi: 10.3892/br.2015.537. Epub 2015 Nov 5. PMID 26870326
- [Background] Sanchez-Vidana DI, Rajwani R, Wong MS. The Use of Omic Technologies Applied to Traditional Chinese Medicine Research. Evid Based Complement Alternat Med. 2017;2017:6359730. doi: 10.1155/2017/6359730. Epub 2017 Jan 31. PMID 28250795
- [Background] Wang XS, Mendoza TR, Gao SZ, Cleeland CS. The Chinese version of the Brief Pain Inventory (BPI-C): its development and use in a study of cancer pain. Pain. 1996 Oct;67(2-3):407-16. doi: 10.1016/0304-3959(96)03147-8. PMID 8951936
- [Background] Yan E, Song J, Liu C, Hong W. A research on syndrome element differentiation based on phenomenology and mathematical method. Chin Med. 2017 Jul 10;12:19. doi: 10.1186/s13020-017-0141-1. eCollection 2017. PMID 28702077
- [Background] Vahedi S. World Health Organization Quality-of-Life Scale (WHOQOL-BREF): Analyses of Their Item Response Theory Properties Based on the Graded Responses Model. Iran J Psychiatry. 2010 Fall;5(4):140-53. PMID 22952508
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Wong W, Lam CL, Wong VT, Yang ZM, Ziea ET, Kwan AK. Validation of the constitution in chinese medicine questionnaire: does the traditional chinese medicine concept of body constitution exist? Evid Based Complement Alternat Med. 2013;2013:481491. doi: 10.1155/2013/481491. Epub 2013 Apr 24. PMID 23710222
- [Background] Karpievitch YV, Polpitiya AD, Anderson GA, Smith RD, Dabney AR. Liquid Chromatography Mass Spectrometry-Based Proteomics: Biological and Technological Aspects. Ann Appl Stat. 2010;4(4):1797-1823. doi: 10.1214/10-AOAS341. PMID 21593992